CLINICAL TRIAL: NCT00732823
Title: A Phase II Randomized Study to Evaluate the Safety of the Compression Test Device Using Intermittent Pneumatic Compression Mode in Subjects With Venous Insufficiency and Oedema
Brief Title: Compression Device Safety Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ConvaTec Inc. (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Professor Dr. med Wolfgang Vanscheidt, Hautarzt Phlebologe Allergologe
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CW-0500-05-U337
Record Dates: First submitted 2008-07-23; First posted 2008-08-12 (Estimated); Last update posted 2008-10-31 (Estimated); Status verified 2008-08

CONDITIONS: Venous Insufficiency
MeSH Terms: conditions — Venous Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Profile A (Placebo Comparator): No device worn
  Interventions: Device: Placebo - No device worn
- Profile B (Active Comparator): Foot 40 mmHg, ankle 40 mmHg, mid-calf 35 mmHg, upper calf 30 mmHg
  Interventions: Device: Prototype device(unnamed)-A battery operated inflatable pneumatic cuffs
- Profile C (Active Comparator): Foot 50 mmHg, ankle 50 mmHg, mid-calf 45 mmHg, upper calf 40 mmHg
  Interventions: Device: Prototype device(unnamed)-A battery operated inflatable pneumatic cuffs
- Profile D (Active Comparator): Foot 60 mmHg, ankle 60 mmHg, mid-calf 55 mmHg, upper calf 50 mmHg
  Interventions: Device: Prototype device(unnamed)-A battery operated inflatable pneumatic cuffs

INTERVENTIONS:
Device: Placebo - No device worn
  Arms: Profile A
Device: Prototype device(unnamed)-A battery operated inflatable pneumatic cuffs
  Arms: Profile B
Device: Prototype device(unnamed)-A battery operated inflatable pneumatic cuffs
  Arms: Profile C
Device: Prototype device(unnamed)-A battery operated inflatable pneumatic cuffs
  Arms: Profile D

SUMMARY:
To evaluate the safety of the Compression Device to subjects with venous insufficiency and oedema.

ELIGIBILITY:
Inclusion Criteria:

* Subjects over 18 years, willing and able to provide written informed consent.
* Subjects able to wear the Amadeus device and follow the requirements of the clinical investigation plan
* Subjects who have an ankle to brachial pressure index (ABPI) of ABPI >0.8
* Subjects with chronic lower limb oedema (i.e. CEAP classification of C3, C4 or C5 1.)
* Subjects who have Chronic Venous Insufficiency (CVI), which has been present for 6 weeks or longer and who have refluxes >0.5 sec in one or more major venous segments, superficial or deep or both (CEAP classification: C3-C5 1.; Ep,s; As,d; Pr).

Exclusion Criteria:

* Subjects with a history of skin sensitivity to any of the components of the study product.
* Subjects who have previously been entered into the study before
* Subjects who have a history of Deep Vein Thrombosis (DVT) within the last 6 months
* Subjects who have an active leg ulcer (i.e. CEAP classification of C6 1).
* Subjects with active cardiac disease or significant history of cardiac disease (including history of myocardial infarction, heart failure, valvular disease, arrhythmia and those with a pacemaker or have previously had a pacemaker).
* Subjects who have initiated treatment or changed the dose within the past month of pharmaceutical agents that reduce clotting e.g. aspirin (except low-dose aspirin), anti-platelets, anti-coagulants and coumarin.
* Subjects who are currently taking pharmaceutical agents that can modify the amount of leg oedema (e.g., diuretics, dihydropyridine calcium channel blockers, phlebotonic drugs, or fluctuating doses of systemic steroids) or have taken these agents within the last 10 days.
* Subjects who are pregnant
* Subjects who have worn compression therapy in the last 48 hours
* Subjects who have leg sizes outside the following range:

  * Ankle 17cm - 32cm
  * Calf 27cm - 47cm
  * Below Knee 29cm - 51cm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2005-07; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
The nature and frequency of adverse events
Distal arterial flow

SECONDARY OUTCOMES:
Volume reduction will be measured by recording limb volume at the start and end of each profile for both legs. The test leg will be compared to baseline and the contralateral leg. Comfort during wear will be recorded on completion of each profile

CONTACTS AND LOCATIONS:
Overall Officials: wolfgang Vanscheidt, Principal Investigator — Facharzt für Dermatologie Phlebologie Allergologie
Locations (1):
- Hautarzt Phlebologe Allergologe, Freiburg im Breisgau, Germany